CLINICAL TRIAL: NCT02456662
Title: A Randomized Controlled Trial of Scheduled Prophylactic Antiemetics for Reduction of Emesis With Doxycycline
Brief Title: Scheduled Prophylactic Antiemetics for Reduction of Emesis With Doxycycline (SPARED) Trial
Acronym: SPARED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Sarah Betstadt, MD, MPH, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RSRB00056271
Record Dates: First submitted 2015-05-26; First posted 2015-05-28 (Estimated); Results first posted 2020-04-16 (Actual); Last update posted 2020-04-16 (Actual); Status verified 2020-04

CONDITIONS: Drug-induced Nausea and Vomiting
MeSH Terms: conditions — Vomiting | interventions — Ondansetron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): 160 Patients will randomly be assigned, using sealed numbered opaque envelopes to receive placebo tablet 30 minutes prior to taking 200mg PO doxycycline
  Interventions: Drug: Placebo
- Ondansetron (Active Comparator): 160 Patients will randomly be assigned, using sealed numbered opaque envelopes to receive 8mg ondansetron tablet 30 minutes prior to taking 200mg PO doxycycline
  Interventions: Drug: Ondansetron

INTERVENTIONS:
Drug: Ondansetron — 8mg PO ondansetron 30 minutes prior to 200mg PO doxycycline
  Other Names: zofran
  Arms: Ondansetron
Drug: Placebo — placebo (identical to study medication- ondansetron) PO 30 minutes prior to 200mg PO doxycycline
  Arms: Placebo

SUMMARY:
Background/Purpose of the Study Doxycycline is an antibiotic used for infection prevention before surgical pregnancy termination, and a side effect of it is nausea/vomiting. The investigators' study explores whether or not taking the anti-emetic ondansetron prior to doxycycline decreases rates of nausea/vomiting. Patients enrolled in the investigators' study will take either ondansetron or a placebo before they take doxycycline to see if ondansetron decreases their nausea/vomiting. Reducing nausea/vomiting may prevent more infections, and decrease the rates of general anesthesia, patient risks and hospital costs. Decreasing nausea/vomiting will also improve patient experience.

Study Design This will be a randomized controlled trial. Data will be collected by administrating surveys and a log where patients will record the timing of their medications and episodes of nausea/vomiting. The primary outcome is nausea/vomiting after taking the anti-emetic/placebo and doxycycline. 400 eligible patients will be enrolled over two years, 200 in the intervention group and 200 in the placebo group.

Rationale for Study Design A randomized controlled trial will be used to determine the effects of the anti-emetic ondansetron on rates of nausea/vomiting.

Subject Characteristics Patients will be pregnant females, 18-45 years old, who are undergoing surgical termination of pregnancy.

Design 1-2 days before the procedure, patients will complete a demographic questionnaire and a survey about symptoms of nausea/vomiting. They will use a log to record symptoms they experience between taking the anti-emetic/placebo and when they present for their procedure. When patients come to the hospital, they will fill out a repeat survey rating their nausea/vomiting.

DETAILED DESCRIPTION:
Scheduled Prophylactic Anti-emetics for Reduction of Emesis with Doxycycline (SPARED) Trial - Study Protocol

Principal Investigator:

Sarah Betstadt, MD MPH Department of Obstetrics & Gynecology University of Rochester Medical Center 601 Elmwood Avenue Rochester, NY 14642-8668 Phone: (585) 276-5367

Co-Investigators:

Amy Harrington, MD

1. PURPOSE OF THE STUDY AND BACKGROUND

   1.1 Purpose of the study The goal of this study is to determine if administering the anti-nausea medication ondansetron prior to doxycycline will decrease the rates of nausea and vomiting in patients taking doxycycline for antibiotic prophylaxis prior to undergoing surgical pregnancy termination.

   1.2 Background The use of prophylactic antibiotics are standard of care to prevent surgical site infections in gynecologic surgery 1. Doxycycline is the recommended antibiotic of choice for surgical pregnancy termination and completion of spontaneous abortion given its effectiveness, low cost, and rare occurrence of allergic reaction 2. Previous studies have shown that a common side effect of doxycycline is nausea and vomiting, with reported rates as high as 30-40% 3. Nausea and vomiting may be reduced by taking the antibiotic with food 4. Doxycycline given on an empty stomach the morning of a surgical pregnancy termination resulted in nausea and vomiting in 50% of patients and this rate was decreased to 15% when it was taken with food the night before surgery 5. It is not known whether the use of scheduled prophylactic anti-emetics prior to doxycycline use would further reduce the rate of associated nausea and vomiting. The goal of the investigators' proposed study is to determine this.

   The investigators' study will be a double blinded randomized controlled trial that will examine whether the use of scheduled prophylactic anti-emetics prior to doxycycline use reduces the incidence of associated nausea and vomiting. Nausea and vomiting is distressing to patients and it affects their perioperative care. It is well documented that minor gynecologic procedures, such as uterine evacuations, can be performed safely with moderate and deep sedation without an endotracheal tube 6. At the investigators' institution, patients experiencing nausea and vomiting prior to a surgical procedure receive general anesthesia with endotracheal intubation, due to their symptoms, not because that would be the preferred route of anesthesia. For minor gynecologic procedures, the time for general anesthesia induction can be as long as the duration of the entire surgical procedure would be without general anesthesia. The use of general anesthesia increases the duration of time in the operating room, which increases the costs of operating room and anesthesia time, as well as recovery time for the patient 7. General anesthesia also poses possible risks such as impairment of cardiovascular function and development of pneumonia 8,9.

   In addition to anesthesia risks and patient discomfort, nausea and vomiting many also affect antibiotic efficacy due to reduced serum levels. Reeves' et al. showed lower serum doxycycline levels in patients with emesis within one hour of doxycycline administration. A serum level greater than 0.8 mg/L has been shown to provide adequate antibiotic prophylaxis. Vomiting after ingestion of doxycycline decreased serum levels by an average of 0.26 mg/L5.

   Reducing the rates of nausea and vomiting in patients undergoing minor gynecologic procedures may increase the efficacy of antibiotic prophylaxis, and decrease the rates of general anesthesia, patient risks and hospital costs. Most importantly, decreased nausea and vomiting will certainly improve patient experience and is clinically relevant because doxycycline is an antibiotic commonly used for many gynecologic procedures.
2. STUDY DESIGN

   2.1 Overview This will be a randomized controlled trial. Data will be collected by asking patients to fill out a demographic questionnaire and a baseline visual analog scale rating their nausea, pain and anxiety at their clinic appointment 1-2 days prior to their procedure. Patients will then take either ondansetron or a placebo 30 minutes prior to taking doxycycline the night before their procedure. They will then fill out a symptom/medication log recording their symptoms from the time that they take the study medication to the time that they present for their procedure. When they present for their procedure, patients will fill out a second identical visual analog scale rating nausea, pain and anxiety. The primary outcome is nausea and vomiting after taking the study drug and doxycycline the night prior to surgery. Doxycycline prophylaxis the night prior to surgery is the current standard of care. Eligible patients will be enrolled over the course of two years. Patients will also have a tube of blood drawn at the time of the procedure so that doxycycline serum levels can be measured.

   2.2 Rationale for Study Design A randomized controlled trial was selected in order to study ondansetron's effect on the rates of nausea and vomiting in the investigators' particular population, so that patient's will not know if they are being given ondansetron or placebo before taking doxycycline. Some potential barriers that are expected in the study include that the patients may not fill out their symptom/medication log as this will be done at home. There are approximately 450 patients undergoing surgical termination of pregnancy at the University of Rochester each year. In order to attain the investigators' goal sample size of 300 patients, the investigators would have to enroll a large portion of the total patients. The primary hypothesis is that the rate of nausea and vomiting in patients undergoing surgical pregnancy termination will be decreased in the group receiving ondansetron versus the group receiving placebo.
3. CHARACERISTICS OF THE RESEARCH POPULATION

   3.1 Subject Characteristics

   3.1.1 Number of Subjects: 300 total subjects are expected to participate in the study. 150 total subjects will be randomized to receive ondansetron, while 150 total subjects will be randomized to receive placebo.

   3.1.2 Gender and Age of Subjects: Patients included in the study will be pregnant females that are ages 18-45 years old.

   3.1.3 Racial and Ethnic Origin: There will be no racial or ethnic restrictions to participation.

   3.1.4 Vulnerable Subjects: The women included in this study will be pregnant, although the study interventions are surveys and the administration of a medication that is both safe in pregnancy and commonly used in pregnancy, ondansetron.

   3.2 Inclusion and Exclusion Criteria

   3.2.1 Inclusion Criteria:
   * Pregnant women seeking care at the University of Rochester's Women's Health Practice Family Planning Clinic
   * Ages 18-45 years old
   * Undergoing second trimester surgical termination of pregnancy
   * Proficient in reading, writing, and comprehending English
   * Able to give informed consent 3.2.2 Exclusion Criteria:
   * Less than 18 years old or older than 45 years old
   * Not proficient in reading, writing, or comprehending English
   * Not able to give informed consent
   * Already taking antiemetics
   * Doxycycline allergy
   * Hyperemesis gravidarum
   * History of gastroparesis or cyclical vomiting
   * Unable to swallow pills

   3.3 Discussion of Subject Population Pregnant women ages 18-45 years old were selected for this study, as they will already be taking doxycycline as the standard of care when they present for abortion care.
4. SUBJECT IDENTIFICATION, RECRUITMENT AND CONSENT

   4.1 Method of Subject Identification and Recruitment Patients presenting for a surgical termination of pregnancy at Women's Health Practice will be offered the opportunity to participate in the study, after they have consented for a pregnancy termination. The investigators offering participation to patients would otherwise have routine contact with these patients, as they will be caring for them regardless of whether or not they participate in the study. If a subject is interested in participating, they will then be screened to determine if they are eligible. Patients will be assigned a random number for the study that will link together their demographic questionnaire, the two visual analog scales, their study drug, and their symptom/medication log.

   4.2 Process of Consent Patients will be consented by either Dr. Sarah Betstadt, Dr. Amy Harrington, research assistant Keelin Abbott, Allison Carletta, NP. The patients will be given a written consent form to sign that will be extensively reviewed with the individual consenting them. The written consents will be stored in a locked filing cabinet, and only Keelin Abbott or Dr. Sarah Betstadt, or Dr. Amy Harrington will be able to access them.
5. METHODS AND STUDY PROCEDURES During their clinic visit 1-2 days before the procedure, patients will fill out a demographic questionnaire regarding their age, race, relationship status, income and education level, pregnancy history, gestational age, and symptoms of nausea and vomiting thus far in the pregnancy. This questionnaire will also include questions regarding cigarette and THC use, as well as any diagnoses of gastroesophageal reflux disease or hyperemesis gravidarum. They will then fill out a baseline visual analog scale rating their nausea, pain and anxiety.

   The patients will then be given a symptom/medication log to take home. The patients will use the log to record symptoms they experience from the time they take the ondansetron or placebo to the time that they present for their procedure. The log will include the timing of the study medication, doxycycline, whether the doxycycline was taken with food (and the time of/type of food if applicable), pain medications, and misoprostol. The log will also include the time of nausea and vomiting, and the severity of the nausea and pain (if applicable).

   When patients present to the hospital for their procedure, research assistant Keelin Abbott, Dr. Amy Harrington, or Dr. Sarah Betstadt will give them a second visual analog scale to fill out which asks them to rate their nausea, pain and anxiety. This scale will be identical to the one they filled out at their clinic visit. This scale will be filled out prior to their procedure.

   Patients will have a tube of blood drawn for a doxycycline serum level upon arrival to the hospital on the day of the procedure.

   5.1 Safety Assessments A comprehensive medical history will be obtained at the patient's clinic visit, and a physical exam will be performed as well to ensure that patients are not only fit and able to undergo their procedure, but also to participate in the study.

   5.2 Assessment of Subject Compliance Compliance with the demographic questionnaire and baseline visual analog scale will be assessed by nature of them both being filled out and turned in in clinic. Compliance with taking the study medication will be assessed by asking the patient if and when they took either the ondansetron or placebo when they present for their procedure. Compliance with completing the symptom/medication log will be assessed by asking the patient to turn in their log when they present for their procedure. Compliance with the second visual analog scale will be ensured by asking the patient to complete it in the hospital before their procedure.

   5.3 Costs to the Subject Subjects will not incur any additional costs by participating in this study.

   5.4 Payment for Participation Patients will not be reimbursed to participate in this study.
6. CONCOMITANT AND DISALLOWED MEDICATIONS As per standard of care (and irrespective of the research study), in addition to doxycycline, patients will take 400 mcg of misoprostol buccally 3 hours before their procedure. It is also standard of care that patients are able to take either Ibuprofen or Tylenol #3 as needed for pain before their procedure. They will also be permitted to take any other medications that they take on a daily basis. None of these medications are part of the research protocol. They will be instructed not to take any antiemetics. The investigators will record any medications that are used.
7. SUBJECT WITHDRAWALS Patients will be withdrawn from the study if they themselves request to do so, or if they fail to take the study medication or the doxycycline. They will not be withdrawn if they fail to complete the demographic questionnaire, the baseline visual analog scale, the symptom/medication log, or the second visual analog scale. In the event that a patient does not complete one of these forms, the investigators' research assistant Keelin Abbott will help her complete them. No additional study activities will be completed prior to subject withdrawal.
8. SAFETY AND REPORTABLE EVENTS 8.1 Adverse Event Definition An adverse event is any symptom, sign, illness, or experience which develops or worsens during the course of the study, whether or not the event is considered related to the study survey.

   8.2 Serious Adverse Event

   A serious adverse event is defined as any adverse medical experience that results in any of the following outcomes:
   * death;
   * is life-threatening;
   * requires inpatient hospitalization or prolongation of existing hospitalization;
   * results in persistent or significant disability/incapacity;
   * is a congenital anomaly/birth defect; or
   * requires medical or surgical intervention to prevent permanent impairment or damage.

   8.3 Recording Adverse Events At each subject visit the site study staff will assess adverse events by recording all voluntary complaints of the subject and by assessment of clinical and laboratory features. At each study visit, the subject should be questioned directly regarding the occurrence of any adverse experience since her last visit.

   All adverse events, whether observed by the Investigator, elicited from or volunteered by the subject, should be documented. Each adverse event will include a brief description of the experience, the time of onset, the time of resolution, the duration and type of experience, the severity, the relationship to the study, contributing factors, and any action taken with respect to the study.

   The recording of adverse events will take place from the time that the subject signs the consent until the subject completes the study (1-2 days after signing the consent) or withdraws from participation.

   8.4 Responsibilities for Reporting Serious Adverse Events All serious adverse experiences that occur during the study period will be recorded. The recording of experiences will occur from the time of signing of the consent until the subject completes the study or withdraws from participation.
9. RISK/BENEFIT ASSESSMENT

   9.1 Risk Category: Greater than minimal risk.

   9.2 Potential Risks Potential risks to subjects include the possibility of an adverse reaction to either ondansetron or placebo, and the potential risk of a patient's greater realization of the nausea and vomiting they are experiencing due to doxycycline. The use of doxycycline is already standard of care.

   9.3 Protection Against Risks The only additional risk may be loss of confidentiality. Study materials will be kept in a locked file cabinet.

   9.4 Potential Benefits to Subjects A potential benefit to subjects participating in this study is a decrease in their nausea and vomiting.

   9.5 Alternatives to Participation Patients who decline to participate in the study will receive the standard of care at the investigators' clinic for termination of pregnancy, which involves the use of doxycycline as a prophylactic antibiotic the night before the procedure, as well as misoprostol the morning of the procedure. They will also be able to take Ibuprofen or Tylenol #3 for pain. They will not fill out any surveys or logs or take the study drug.
10. CONFIDENTIALITY OF DATA AND INFORMATION STORAGE 10.1 Subject data will be identified in the research data set by random unique identifiable code. Research assistant Keelin Abbott will maintain the code to that information and it will be used to re-identify patients when they present for their procedure, in order to link together their demographic questionnaire, the two visual analog scales, their study medication, and the symptom/medication log. The research data will be secured in a locked filing cabinet during the study. No identifying information will be included in the research database except for the subject's ID number, any identifying information will be kept separately from the research database. Research files will be locked up when they are unsupervised, and only Keelin Abbott, Dr. Sarah Betsadt, or Dr. Amy Harrington will be able to access the files.
11. RESEARCH INFORMATION IN MEDICAL RECORDS No research data will be included in the subject's medical record.
12. DATA ANALYSIS AND MONITORING 12.1 Sample Size Determination Based on Reeves' study as well as anecdotal data from the investigators' clinic population, the investigators expect vomiting to occur in approximately 30% of the investigators' patients who take their doxycycline the night before their procedure. To have 80% power to detect a 50% decrease in nausea and vomiting, the investigators will need 122 patients in each arm of the study. In order to account for subject withdrawal or non-compliance, the investigators intend to enroll 150 patients in each arm of the study.

12.2 Planned Statistical Analysis Our primary outcome of vomiting, will be analyzed using chi-square analysis. All dichotomous outcomes will be analyzed using chi-square analysis. Continuous variables will be examined using t-tests. If demographic variables are found to be confounders with significance, they will be placed into a logistic regression model. SPSS software will be used for statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women seeking care at the University of Rochester's Women's Health Practice Family Planning Clinic
* Undergoing second trimester surgical termination of pregnancy
* Proficient in reading, writing, and comprehending English
* Able to give informed consent

Exclusion Criteria:

* Not proficient in reading, writing, or comprehending English
* Not able to give informed consent
* Already taking antiemetics
* Doxycycline allergy
* Hyperemesis gravidarum
* History of gastroparesis or cyclical vomiting
* Unable to swallow pills

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 319 (Actual)
Dates: Start 2015-10-07; Primary Completion 2019-04-03 (Actual); Study Completion 2019-04-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah J Betstadt, MD, MPH, Principal Investigator — University of Rochester
Locations (1):
- Lattimore Women's Health Practice, Rochester, New York, United States

REFERENCES:
- [Background] Sawaya GF, Grady D, Kerlikowske K, Grimes DA. Antibiotics at the time of induced abortion: the case for universal prophylaxis based on a meta-analysis. Obstet Gynecol. 1996 May;87(5 Pt 2):884-90. PMID 8677129
- [Background] Bryant SG, Fisher S, Kluge RM. Increased frequency of doxycycline side effects. Pharmacotherapy. 1987;7(4):125-9. doi: 10.1002/j.1875-9114.1987.tb04037.x. PMID 3684731
- [Background] Risser W. Side effects of doxycycline in adolescents treated for pelvic inflammatory disease. J Pediatr Adolesc Gynecol. 2011 Jun;24(3):e87. doi: 10.1016/j.jpag.2011.02.010. No abstract available. PMID 21601804
- [Background] Reeves MF, Lohr PA, Hayes JL, Harwood BJ, Creinin MD. Doxycycline serum levels at the time of dilation and evacuation with two dosing regimens. Contraception. 2009 Feb;79(2):129-33. doi: 10.1016/j.contraception.2008.09.006. Epub 2008 Nov 13. PMID 19135570
- [Background] Dean G, Jacobs AR, Goldstein RC, Gevirtz CM, Paul ME. The safety of deep sedation without intubation for abortion in the outpatient setting. J Clin Anesth. 2011 Sep;23(6):437-42. doi: 10.1016/j.jclinane.2011.05.001. Epub 2011 Aug 9. PMID 21831622
- [Background] Brooks DM, Hand WR Jr. A cost analysis: general endotracheal versus regional versus monitored anesthesia care. Mil Med. 1999 Apr;164(4):303-5. PMID 10226461
- [Background] ACOG practice bulletin No. 104: antibiotic prophylaxis for gynecologic procedures. Obstet Gynecol. 2009 May;113(5):1180-1189. doi: 10.1097/AOG.0b013e3181a6d011. No abstract available. PMID 19384149

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 757 participants were screened. 438 were excluded because they were not eligible or declined to participate. 319 were randomized to either placebo or Ondansetron.
Period: Overall Study
Arm/Group | Placebo | Ondansetron
Started | 159 | 160
Completed | 157 | 159
Not Completed | 2 | 1
Not completed — Lost to Follow-up | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Ondansetron | Total
Number analyzed (Participants) | 159 | 160 | 319
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Age data was not collected on one participant in the placebo arm.
  years
    number analyzed (Participants) | 158 | 160 | 318
    (all) | 26.0 (5.8) | 26.4 (5.8) | 26.2 (5.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 159 | 160 | 319
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 12 | 27
  Not Hispanic or Latino | 141 | 147 | 288
  Unknown or Not Reported | 3 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 3 | 5
  Asian | 0 | 3 | 3
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 58 | 57 | 115
  White | 79 | 81 | 160
  More than one race | 13 | 11 | 24
  Unknown or Not Reported | 6 | 4 | 10
Region of Enrollment [Number; unit: participants]
  United States | 159 | 160 | 319

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Symptoms
Description: Number of participants experiencing symptoms (vomiting or nausea+vomiting) at the time of or after doxycycline
Time Frame: 24 hours
Population: This was an intent to treat analysis so all participants were included.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ondansetron
Number analyzed (Participants) | 159 | 160
Participants | 45 | 19
Statistical Analysis 1: Comparison: Placebo vs Ondansetron; Test type: Superiority — Based on previous work as well as anecdotal data from our clinic population, we expect vomiting to occur in approximately 30% of our patients who take their doxycycline the night before their procedure. To have 80% power to detect a 50% decrease in nausea and vomiting, we will need 122 patients in each arm of the study; p = 0.00, Chi-squared

ADVERSE EVENTS:
Time Frame: 24 hours
Arm/Group | Placebo | Ondansetron
All-Cause Mortality (participants affected / at risk) | 0/159 | 0/160
Serious Adverse Events (participants affected / at risk) | 0/159 | 0/160
Other Adverse Events (participants affected / at risk) | 0/159 | 0/160

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-06-22): https://cdn.clinicaltrials.gov/large-docs/62/NCT02456662/Prot_SAP_000.pdf
  • Informed Consent Form (2018-07-23): https://cdn.clinicaltrials.gov/large-docs/62/NCT02456662/ICF_001.pdf